CLINICAL TRIAL: NCT06290713
Title: Vasodilators and Exercise as Adjuvant Therapy for Duchenne Muscular Dystrophy (VASO-REx Study)
Brief Title: Vasodilator and Exercise Study for DMD (VASO-REx)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB202301491; 1R21AR079755-01 (NIH); PRO00050023 (Other: UFIRST)
Record Dates: First submitted 2024-02-09; First posted 2024-03-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-02

CONDITIONS: Duchenne Muscular Dystrophy; Duchenne Disease; Muscular Dystrophy; Muscular Dystrophy in Children; Vasodilation; Exercise; DMD
Keywords: DMD; Tadalafil; Drug and Exercise Intervention; Treatment Strategy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Tabes Dorsalis; Muscular Dystrophies; Aneurysm; Motor Activity | interventions — Tadalafil; Exercise

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive interventions based on their completion and results of Aim 1 (responsiveness to study drug). If participants are found to be Tadalafil-responsive after one dose, they will be included in Aim 2 of the study and will be asked to participate in the double-blinded, randomized, placebo-controlled longitudinal medication & exercise 6-month study program.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tadalafil and Exercise Arm (Experimental): Participants receive tadalafil weight-dependent dosage to take daily for 6 months (26 weeks).
  Interventions: Drug: Tadalafil; Other: Exercise Training
- Placebo and Exercise Arm (Placebo Comparator): Participants receive a tadalafil placebo tablet matching the tadalafil weight-dependent dosage to take daily for 6 months (26 weeks).
  Interventions: Drug: Placebo; Other: Exercise Training

INTERVENTIONS:
Drug: Tadalafil — Patients will be given either the intervention medication or a placebo (double-blinded, randomized trial) and will be asked to take the medication every day for 6 months in conjunction with weekly exercise sessions.
  Arms: Tadalafil and Exercise Arm
Drug: Placebo — Patients will be given either the intervention medication or a placebo (double-blinded, randomized trial) and will be asked to take the medication every day for 6 months in conjunction with weekly exercise sessions.
  Arms: Placebo and Exercise Arm
Other: Exercise Training — The home-based cycling exercise training program is designed to improve muscle strength and endurance. Participants will engage in individualized exercise sessions up to four times per week, lasting up to 40 minutes each. Live video and heart rate monitoring will ensure proper exercise performance and allow for adjustments to the program throughout the study. The participants will receive the exercise equipment for use at home.

SUMMARY:
Examining two strategies as potential adjuvant therapies for Duchenne muscular dystrophy (DMD); aerobic exercise training (to induce adaptations in skeletal muscle and improve cardiovascular health) and tadalafil, an FDA-approved vasodilator (to optimize blood flow and muscle perfusion which is impaired and often overlooked in DMD). Target: improved muscle function, vascular health, and DMD treatment.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is characterized by rapid muscle deterioration, mitochondrial and vascular impairments, resulting in premature loss of ambulation and mortality. Disease-modifying therapeutics are emerging and although they are expected to improve muscle function and daily activity in boys with DMD, most are not designed to correct the vascular impairment. This impairment is due to the lack of restoration of neuronal nitric oxide synthase signaling, which is crucial for vasodilation during and after exercise. The investigators believe limitations in study design were responsible for the lack of efficacy. Therefore, this study combines tadalafil with aerobic exercise to necessitate increased blood flow and activate the drug.

This Exploratory Clinical Trial will assess two potential adjuvant therapies for ambulatory boys with DMD (6 years and older): 1) aerobic exercise training and 2) tadalafil, an FDA-approved vasodilator drug. Preclinical and clinical data, including recent findings from the principal investigator's lab, support the use of these strategies and their potential to benefit muscle perfusion, fatigue, and quality of life.

The study will first test for drug responsiveness (increase in muscle oxygenation) after a single dose. Drug-responsive boys with DMD will be randomized to a 6-month intervention of daily tadalafil or placebo, combined with structured cycle exercise training. Participants will receive exercise-related equipment for use at home and be monitored by the research team via video. The study will quantify the intervention's impact on vascular impairment, muscle pathophysiology (inflammation, fat accumulation, mitochondrial dysfunction), exertional fatigue, and cycling performance.

Our findings are expected to yield:

1. Criteria to identify DMD patients most likely to benefit from tadalafil as adjuvant therapy.
2. Evidence of a powerful synergy between drug impact and exercise training in DMD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD confirmed by genetic report
* Minimum entry age of 6.0 years old
* Ambulatory
* On stable glucocorticoid regimen (for > 3 months)

Exclusion Criteria:

* Contraindication to a Magnetic resonance Imaging examination (e.g. severe claustrophobia, magnetic implants, unable/unwilling to perform test)
* Presence of unstable medical problems, including severe cardiomyopathy, left ventricular ejection fraction <45%, cardiac conduction abnormalities as evidenced on ECG, uncontrolled seizure disorder, uncontrolled hypo or hypertension
* Presence of a secondary condition that impacts muscle function or muscle metabolism (e.g., myasthenia gravis, endocrine disorder, mitochondrial disease)
* Presence of a secondary condition leading to developmental delay or impaired motor control (e.g., cerebral palsy) or previous history of unprovoked rhabdomyolysis
* Contraindications to phosphodiesterase 5 inhibitors (use of nitrates, alpha-adrenergic blockers, other phosphodiesterase 5 inhibitors) or other medications known to modulate blood flow or muscle metabolism
* Participation in currently approved FDA trials or other investigational clinical trials during the period of the study

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Duchenne Muscular Dystrophy is an X-linked disorder, and therefore predominantly in males. As a result, the principal investigator is limiting the children study participants to males.
Enrollment: 50 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Vascular responsiveness after muscle contraction to a single dose of tadalafil. | up to 4 weeks after the completion of Visits 1 and 2 of Aim 1.
  Responsiveness will be determined by an increase in post-contractile muscle oxygenation using MRI-Blood Oxygen Level Dependent (BOLD) responses after dosing compared to before. Study participants demonstrating an increase (>50%) in post-contractile BOLD after tadalafil will be enrolled into Aim 2 of this study.
Cycling time to fatigue | Baseline and 6 month follow-up visits of Aim 2.
  The study will assess the impact of tadalafil on exercise performance and fatigue resistance compared to placebo. Participants will undergo a maximal effort cycling test before and after the intervention period. The time it takes for participants to reach exhaustion (TTE) will be recorded as the primary outcome measure.
  Measurement: Time to exhaustion (TTE) during a maximal effort cycling test on a recumbent, stationary ergometer. This test will quantify fatigue resistance by measuring the duration participants can sustain maximal effort cycling.

SECONDARY OUTCOMES:
Quadriceps muscle Fat Fraction | Aim 1 and Aim 2 (baseline and 6 month follow-up)
  This outcome serves as a measure of disease severity. This measure is a sensitive and reproducible biomarker of DMD muscle pathology.
Metabolic recovery | Through study completion, an average of 3 years.
  The rate of phosphocreatine resynthesis after leg exercise will be quantified and serves as index of skeletal muscle mitochondrial oxidative capacity. (Part of Aim 2 of the study).
cardiopulmonary exercise testing (CPET) - Peak aerobic capacity (VO2max) | Through study completion, an average of 3 years.
  Patients will undergo cycling exercise at submaximal and peak workloads to quantify peak aerobic capacity, ventilation.
  Peak Oxygen Uptake (VO2max): This measure quantifies the maximum amount of oxygen the body can utilize during exercise, assessed through maximal cycling effort in a CPET. It serves as a primary indicator of overall cardiovascular and aerobic fitness.
  Peak aerobic capacity: VO2max reflects the maximum oxygen utilization capacity, indicating overall cardiovascular fitness.
cardiopulmonary exercise testing (CPET) - Minute Ventilation (VE) | Through study completion, an average of 3 years.
  Minute Ventilation (VE): This measure reflects the total volume of air breathed per minute during exercise, assessed throughout the CPET. Evaluating VE at various workloads provides insights into respiratory efficiency and potential limitations during exercise.
  Respiratory efficiency: VE and VE/VO2 assess how well the body utilizes oxygen during exercise, revealing potential respiratory limitations.
cardiopulmonary exercise testing (CPET) - Ventilatory Equivalent for Oxygen (VE/VO2) | Through study completion, an average of 3 years.
  Ventilatory Equivalent for Oxygen (VE/VO2): This ratio compares ventilation to oxygen uptake, calculated throughout the CPET. It indicates the efficiency of oxygen utilization during exercise and potential respiratory limitations.
  Respiratory efficiency: VE and VE/VO2 assess how well the body utilizes oxygen during exercise, revealing potential respiratory limitations.
cardiopulmonary exercise testing (CPET) - Gas Exchange Threshold (GET) | Through study completion, an average of 3 years.
  Gas Exchange Threshold (GET): This point during exercise marks the transition from predominantly aerobic to anaerobic metabolism, identified through changes in blood lactate levels and other CPET parameters. Analyzing GET helps assess exercise tolerance and potential for improvement.
  Exercise tolerance and fatigue: GET and W at AT pinpoint the intensity at which fatigue and performance decline become significant, offering insights into exercise limitations and potential for improvement.
cardiopulmonary exercise testing (CPET) - Workload at Anaerobic Threshold (W at AT) | Through study completion, an average of 3 years.
  Workload at Anaerobic Threshold (W at AT): This measure, derived from the CPET, quantifies the power output at which anaerobic metabolism significantly contributes to energy production. It reflects exercise intensity at which fatigue and performance decline become prominent.
  Exercise tolerance and fatigue: GET and W at AT pinpoint the intensity at which fatigue and performance decline become significant, offering insights into exercise limitations and potential for improvement.
The 100-meter timed test (100m) | Through study completion, an average of 3 years.
  The 100m is a fixed distance test of maximal performance and will be completed according to published guidelines.
the North Star Ambulatory Assessment (NSAA) | Through study completion, an average of 3 years.
  The North Star Ambulatory Assessment (NSAA) is a 17-item rating scale that is used to measure physical function and motor abilities in ambulatory boys with DMD and is increasingly being used in clinical trials as an overall measure of physical function.
The 4-stair climb | Through study completion, an average of 3 years.
  The time to ascend 4-stairs is a strength-measure. The patient is instructed to climb four standard steps (six inches in height each) with two handrails as fast as safely possible, using the rails if needed.
The Physical activity questionnaire (PAQ-C) | Through study completion, an average of 3 years.
  The PAQ-C is a self-administered, 7-day recall instrument developed to assess general levels of physical activity throughout the elementary school year for students in grades 4 to 8 and approximately 8 to 14 years, with high validity. Although reliability is considered to be moderate, other physical activity questionnaires are less reliable. Results will be correlated with indices of disease severity and tadalafil responsiveness.
Pulmonary function testing - vital capacity (FVC) | Through study completion, an average of 3 years.
  Measurement: FVC, measured using a standard spirometer according to American Thoracic Society guidelines. This is the maximum amount of air an individual can forcefully exhale after a full inhalation.
  Significance: FVC reflects the total lung capacity and is a key indicator of overall lung volume and function. It can help identify restrictive lung diseases, where lung volume is limited, and track respiratory health changes over time.
Pulmonary function testing - forced expiratory volume in 1 second (FEV1) | Through study completion, an average of 3 years.
  Measurement: FEV1, measured using a standard spirometer according to American Thoracic Society guidelines. This is the amount of air forcefully exhaled in the first second of a maximal exhalation after a full inhalation.
  Significance: FEV1 reflects the efficiency of airflow from the lungs and is sensitive to obstructive lung diseases, like asthma and Chronic Obstructive Pulmonary Disease (COPD), where airflow is impaired.
Neurology Quality of Life (NeuroQoL) pediatric lower extremity function | Through study completion, an average of 3 years.
  Questionnaire used to measure patient-reported outcomes of intervention impact.
Patient Reported Outcomes Measurement Information System (PROMIS) pediatric fatigue | Through study completion, an average of 3 years.
  Questionnaire used to measure patient-reported outcomes of intervention impact.
PROMIS parent proxy for physical activity | Through study completion, an average of 3 years.
  Questionnaire used to measure patient's parent-reported outcomes of intervention impact.
PROMIS pediatric physical activity | Through study completion, an average of 3 years.
  Questionnaire used to measure patient's parent-reported outcomes of intervention impact.
Physical Activity Monitoring - Daily Step Rate | Through study completion, an average of 3 years.
  Measurement: Total number of steps taken per day, assessed using the Actigraph activity monitor.
Physical Activity Monitoring - Time in Low-Level Activity | Through study completion, an average of 3 years.
  Measurement: Total time spent in low-intensity physical activity per day, as defined by Actigraph criteria.
Physical Activity Monitoring - Time in Moderate-Level Activity | Through study completion, an average of 3 years.
  Measurement: Total time spent in moderate-intensity physical activity per day, as defined by Actigraph criteria.
Physical Activity Monitoring - Time in High-Level Activity | Through study completion, an average of 3 years.
  Measurement: Total time spent in high-intensity physical activity per day, as defined by Actigraph criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Taivassalo, Ph.D., Principal Investigator — University of Florida, College of Medicine, Department of Physiology and Aging
Locations (1):
- University of Florida Clinical and Translational Research Building, Gainesville, Florida, United States

REFERENCES:
- [Background] Lopez C, Taivassalo T, Berru MG, Saavedra A, Rasmussen HC, Batra A, Arora H, Roetzheim AM, Walter GA, Vandenborne K, Forbes SC. Postcontractile blood oxygenation level-dependent (BOLD) response in Duchenne muscular dystrophy. J Appl Physiol (1985). 2021 Jul 1;131(1):83-94. doi: 10.1152/japplphysiol.00634.2020. Epub 2021 May 20. PMID 34013753
- [Background] Mendell JR, Sahenk Z, Lehman K, Nease C, Lowes LP, Miller NF, Iammarino MA, Alfano LN, Nicholl A, Al-Zaidy S, Lewis S, Church K, Shell R, Cripe LH, Potter RA, Griffin DA, Pozsgai E, Dugar A, Hogan M, Rodino-Klapac LR. Assessment of Systemic Delivery of rAAVrh74.MHCK7.micro-dystrophin in Children With Duchenne Muscular Dystrophy: A Nonrandomized Controlled Trial. JAMA Neurol. 2020 Sep 1;77(9):1122-1131. doi: 10.1001/jamaneurol.2020.1484. PMID 32539076
- [Background] Harper SQ. Molecular dissection of dystrophin identifies the docking site for nNOS. Proc Natl Acad Sci U S A. 2013 Jan 8;110(2):387-8. doi: 10.1073/pnas.1220256110. Epub 2012 Dec 31. No abstract available. PMID 23277550
- [Background] Duan D. Systemic AAV Micro-dystrophin Gene Therapy for Duchenne Muscular Dystrophy. Mol Ther. 2018 Oct 3;26(10):2337-2356. doi: 10.1016/j.ymthe.2018.07.011. Epub 2018 Jul 17. PMID 30093306
- [Background] Percival JM, Adamo CM, Beavo JA, Froehner SC. Evaluation of the therapeutic utility of phosphodiesterase 5A inhibition in the mdx mouse model of duchenne muscular dystrophy. Handb Exp Pharmacol. 2011;(204):323-44. doi: 10.1007/978-3-642-17969-3_14. PMID 21695647
- [Background] Thomas GD. Functional muscle ischemia in Duchenne and Becker muscular dystrophy. Front Physiol. 2013 Dec 18;4:381. doi: 10.3389/fphys.2013.00381. PMID 24391598
- [Background] Kobayashi YM, Rader EP, Crawford RW, Iyengar NK, Thedens DR, Faulkner JA, Parikh SV, Weiss RM, Chamberlain JS, Moore SA, Campbell KP. Sarcolemma-localized nNOS is required to maintain activity after mild exercise. Nature. 2008 Nov 27;456(7221):511-5. doi: 10.1038/nature07414. Epub 2008 Oct 26. PMID 18953332
- [Background] Sheffield-Moore M, Wiktorowicz JE, Soman KV, Danesi CP, Kinsky MP, Dillon EL, Randolph KM, Casperson SL, Gore DC, Horstman AM, Lynch JP, Doucet BM, Mettler JA, Ryder JW, Ploutz-Snyder LL, Hsu JW, Jahoor F, Jennings K, White GR, McCammon SD, Durham WJ. Sildenafil increases muscle protein synthesis and reduces muscle fatigue. Clin Transl Sci. 2013 Dec;6(6):463-8. doi: 10.1111/cts.12121. Epub 2013 Oct 29. PMID 24330691
- [Background] Nelson MD, Rader F, Tang X, Tavyev J, Nelson SF, Miceli MC, Elashoff RM, Sweeney HL, Victor RG. PDE5 inhibition alleviates functional muscle ischemia in boys with Duchenne muscular dystrophy. Neurology. 2014 Jun 10;82(23):2085-91. doi: 10.1212/WNL.0000000000000498. Epub 2014 May 7. PMID 24808022
- [Background] Victor RG, Sweeney HL, Finkel R, McDonald CM, Byrne B, Eagle M, Goemans N, Vandenborne K, Dubrovsky AL, Topaloglu H, Miceli MC, Furlong P, Landry J, Elashoff R, Cox D; Tadalafil DMD Study Group. A phase 3 randomized placebo-controlled trial of tadalafil for Duchenne muscular dystrophy. Neurology. 2017 Oct 24;89(17):1811-1820. doi: 10.1212/WNL.0000000000004570. Epub 2017 Sep 29. PMID 28972192
- [Background] Hoffman EP. Pharmacotherapy of Duchenne Muscular Dystrophy. Handb Exp Pharmacol. 2020;261:25-37. doi: 10.1007/164_2019_256. PMID 31375923
- [Background] Mah JK. An Overview of Recent Therapeutics Advances for Duchenne Muscular Dystrophy. Methods Mol Biol. 2018;1687:3-17. doi: 10.1007/978-1-4939-7374-3_1. PMID 29067652
- [Background] Verhaart IEC, Aartsma-Rus A. Therapeutic developments for Duchenne muscular dystrophy. Nat Rev Neurol. 2019 Jul;15(7):373-386. doi: 10.1038/s41582-019-0203-3. PMID 31147635
- [Background] Ramos JN, Hollinger K, Bengtsson NE, Allen JM, Hauschka SD, Chamberlain JS. Development of Novel Micro-dystrophins with Enhanced Functionality. Mol Ther. 2019 Mar 6;27(3):623-635. doi: 10.1016/j.ymthe.2019.01.002. Epub 2019 Feb 1. PMID 30718090
- [Background] Lai Y, Thomas GD, Yue Y, Yang HT, Li D, Long C, Judge L, Bostick B, Chamberlain JS, Terjung RL, Duan D. Dystrophins carrying spectrin-like repeats 16 and 17 anchor nNOS to the sarcolemma and enhance exercise performance in a mouse model of muscular dystrophy. J Clin Invest. 2009 Mar;119(3):624-35. doi: 10.1172/JCI36612. Epub 2009 Feb 23. PMID 19229108
- [Background] Khan N, Eliopoulos H, Han L, Kinane TB, Lowes LP, Mendell JR, Gordish-Dressman H, Henricson EK, McDonald CM; Eteplirsen Investigators and the CINRG DNHS Investigators. Eteplirsen Treatment Attenuates Respiratory Decline in Ambulatory and Non-Ambulatory Patients with Duchenne Muscular Dystrophy. J Neuromuscul Dis. 2019;6(2):213-225. doi: 10.3233/JND-180351. PMID 30856119
- [Background] Charleston JS, Schnell FJ, Dworzak J, Donoghue C, Lewis S, Chen L, Young GD, Milici AJ, Voss J, DeAlwis U, Wentworth B, Rodino-Klapac LR, Sahenk Z, Frank D, Mendell JR. Eteplirsen treatment for Duchenne muscular dystrophy: Exon skipping and dystrophin production. Neurology. 2018 Jun 12;90(24):e2146-e2154. doi: 10.1212/WNL.0000000000005680. Epub 2018 May 11. PMID 29752304
- [Background] Mendell JR, Engel WK, Derrer EC. Duchenne muscular dystrophy: functional ischemia reproduces its characteristic lesions. Science. 1971 Jun 11;172(3988):1143-5. doi: 10.1126/science.172.3988.1143. PMID 5574520
- [Background] Rando TA. Role of nitric oxide in the pathogenesis of muscular dystrophies: a "two hit" hypothesis of the cause of muscle necrosis. Microsc Res Tech. 2001 Nov 15;55(4):223-35. doi: 10.1002/jemt.1172. PMID 11748861
- [Background] Dietz AR, Connolly A, Dori A, Zaidman CM. Intramuscular blood flow in Duchenne and Becker Muscular Dystrophy: Quantitative power Doppler sonography relates to disease severity. Clin Neurophysiol. 2020 Jan;131(1):1-5. doi: 10.1016/j.clinph.2019.09.023. Epub 2019 Nov 4. PMID 31751835
- [Background] Mutlu A, Alkan H, Firat T, Karaduman AA, Yilmaz OT. How do physical capacity, fatigue and performance differ in children with duchenne muscular dystrophy compared with their healthy peers? Neurosciences (Riyadh). 2018 Jan;23(1):39-45. doi: 10.17712/nsj.2018.1.20170242. PMID 29455220
- [Background] Gentil C, Leturcq F, Ben Yaou R, Kaplan JC, Laforet P, Penisson-Besnier I, Espil-Taris C, Voit T, Garcia L, Pietri-Rouxel F. Variable phenotype of del45-55 Becker patients correlated with nNOSmu mislocalization and RYR1 hypernitrosylation. Hum Mol Genet. 2012 Aug 1;21(15):3449-60. doi: 10.1093/hmg/dds176. Epub 2012 May 15. PMID 22589245
- [Background] Nelson MD, Rosenberry R, Barresi R, Tsimerinov EI, Rader F, Tang X, Mason O, Schwartz A, Stabler T, Shidban S, Mobaligh N, Hogan S, Elashoff R, Allen JD, Victor RG. Sodium nitrate alleviates functional muscle ischaemia in patients with Becker muscular dystrophy. J Physiol. 2015 Dec 1;593(23):5183-200. doi: 10.1113/JP271252. Epub 2015 Nov 2. PMID 26437761
- [Background] Boehler JF, Ricotti V, Gonzalez JP, Soustek-Kramer M, Such L, Brown KJ, Schneider JS, Morris CA. Membrane recruitment of nNOSmicro in microdystrophin gene transfer to enhance durability. Neuromuscul Disord. 2019 Oct;29(10):735-741. doi: 10.1016/j.nmd.2019.08.009. Epub 2019 Aug 23. PMID 31521486
- [Background] Balke JE, Zhang L, Percival JM. Neuronal nitric oxide synthase (nNOS) splice variant function: Insights into nitric oxide signaling from skeletal muscle. Nitric Oxide. 2019 Jan 1;82:35-47. doi: 10.1016/j.niox.2018.11.004. Epub 2018 Nov 29. PMID 30503614
- [Background] Asai A, Sahani N, Kaneki M, Ouchi Y, Martyn JA, Yasuhara SE. Primary role of functional ischemia, quantitative evidence for the two-hit mechanism, and phosphodiesterase-5 inhibitor therapy in mouse muscular dystrophy. PLoS One. 2007 Aug 29;2(8):e806. doi: 10.1371/journal.pone.0000806. PMID 17726536
- [Background] De Arcangelis V, Strimpakos G, Gabanella F, Corbi N, Luvisetto S, Magrelli A, Onori A, Passananti C, Pisani C, Rome S, Severini C, Naro F, Mattei E, Di Certo MG, Monaco L. Pathways Implicated in Tadalafil Amelioration of Duchenne Muscular Dystrophy. J Cell Physiol. 2016 Jan;231(1):224-32. doi: 10.1002/jcp.25075. PMID 26097015
- [Background] Webster C, Silberstein L, Hays AP, Blau HM. Fast muscle fibers are preferentially affected in Duchenne muscular dystrophy. Cell. 1988 Feb 26;52(4):503-13. doi: 10.1016/0092-8674(88)90463-1. PMID 3342447
- [Background] Batra A, Vohra RS, Chrzanowski SM, Hammers DW, Lott DJ, Vandenborne K, Walter GA, Forbes SC. Effects of PDE5 inhibition on dystrophic muscle following an acute bout of downhill running and endurance training. J Appl Physiol (1985). 2019 Jun 1;126(6):1737-1745. doi: 10.1152/japplphysiol.00664.2018. Epub 2019 Apr 4. PMID 30946638
- [Background] McDonald CM, Henricson EK, Abresch RT, Florence JM, Eagle M, Gappmaier E, Glanzman AM; PTC124-GD-007-DMD Study Group; Spiegel R, Barth J, Elfring G, Reha A, Peltz S. The 6-minute walk test and other endpoints in Duchenne muscular dystrophy: longitudinal natural history observations over 48 weeks from a multicenter study. Muscle Nerve. 2013 Sep;48(3):343-56. doi: 10.1002/mus.23902. Epub 2013 Jun 26. PMID 23681930
- [Background] Hoffman EP, Connor EM. Orphan drug development in muscular dystrophy: update on two large clinical trials of dystrophin rescue therapies. Discov Med. 2013 Nov;16(89):233-9. PMID 24229740
- [Background] Fowler EG, Staudt LA, Heberer KR, Sienko SE, Buckon CE, Bagley AM, Sussman MD, McDonald CM. Longitudinal community walking activity in Duchenne muscular dystrophy. Muscle Nerve. 2018 Mar;57(3):401-406. doi: 10.1002/mus.25743. Epub 2017 Jul 28. PMID 28692198
- [Background] McDonald CM, Henricson EK, Abresch RT, Han JJ, Escolar DM, Florence JM, Duong T, Arrieta A, Clemens PR, Hoffman EP, Cnaan A; Cinrg Investigators. The cooperative international neuromuscular research group Duchenne natural history study--a longitudinal investigation in the era of glucocorticoid therapy: design of protocol and the methods used. Muscle Nerve. 2013 Jul;48(1):32-54. doi: 10.1002/mus.23807. Epub 2013 May 16. PMID 23677550
- [Background] Bloom TJ. Age-related alterations in cyclic nucleotide phosphodiesterase activity in dystrophic mouse leg muscle. Can J Physiol Pharmacol. 2005 Nov;83(11):1055-60. doi: 10.1139/y05-085. PMID 16391714
- [Background] Witting N, Kruuse C, Nyhuus B, Prahm KP, Citirak G, Lundgaard SJ, von Huth S, Vejlstrup N, Lindberg U, Krag TO, Vissing J. Effect of sildenafil on skeletal and cardiac muscle in Becker muscular dystrophy. Ann Neurol. 2014 Oct;76(4):550-7. doi: 10.1002/ana.24216. Epub 2014 Jul 15. PMID 25042931
- [Background] Leung DG, Herzka DA, Thompson WR, He B, Bibat G, Tennekoon G, Russell SD, Schuleri KH, Lardo AC, Kass DA, Thompson RE, Judge DP, Wagner KR. Sildenafil does not improve cardiomyopathy in Duchenne/Becker muscular dystrophy. Ann Neurol. 2014 Oct;76(4):541-9. doi: 10.1002/ana.24214. Epub 2014 Jul 10. PMID 25042693
- [Background] Zhang L, Zhang Z, Zhang RL, Cui Y, LaPointe MC, Silver B, Chopp M. Tadalafil, a long-acting type 5 phosphodiesterase isoenzyme inhibitor, improves neurological functional recovery in a rat model of embolic stroke. Brain Res. 2006 Nov 6;1118(1):192-8. doi: 10.1016/j.brainres.2006.08.028. Epub 2006 Sep 7. PMID 16959227
- [Background] Ledermann HP, Schulte AC, Heidecker HG, Aschwanden M, Jager KA, Scheffler K, Steinbrich W, Bilecen D. Blood oxygenation level-dependent magnetic resonance imaging of the skeletal muscle in patients with peripheral arterial occlusive disease. Circulation. 2006 Jun 27;113(25):2929-35. doi: 10.1161/CIRCULATIONAHA.105.605717. Epub 2006 Jun 19. PMID 16785340
- [Background] Slade JM, Towse TF, Gossain VV, Meyer RA. Peripheral microvascular response to muscle contraction is unaltered by early diabetes but decreases with age. J Appl Physiol (1985). 2011 Nov;111(5):1361-71. doi: 10.1152/japplphysiol.00009.2011. Epub 2011 Jul 28. PMID 21799123
- [Background] Towse TF, Slade JM, Ambrose JA, DeLano MC, Meyer RA. Quantitative analysis of the postcontractile blood-oxygenation-level-dependent (BOLD) effect in skeletal muscle. J Appl Physiol (1985). 2011 Jul;111(1):27-39. doi: 10.1152/japplphysiol.01054.2009. Epub 2011 Feb 17. PMID 21330621
- [Background] Forbes SC, Walter GA, Rooney WD, Wang DJ, DeVos S, Pollaro J, Triplett W, Lott DJ, Willcocks RJ, Senesac C, Daniels MJ, Byrne BJ, Russman B, Finkel RS, Meyer JS, Sweeney HL, Vandenborne K. Skeletal muscles of ambulant children with Duchenne muscular dystrophy: validation of multicenter study of evaluation with MR imaging and MR spectroscopy. Radiology. 2013 Oct;269(1):198-207. doi: 10.1148/radiol.13121948. Epub 2013 May 21. PMID 23696684
- [Background] Willcocks RJ, Rooney WD, Triplett WT, Forbes SC, Lott DJ, Senesac CR, Daniels MJ, Wang DJ, Harrington AT, Tennekoon GI, Russman BS, Finanger EL, Byrne BJ, Finkel RS, Walter GA, Sweeney HL, Vandenborne K. Multicenter prospective longitudinal study of magnetic resonance biomarkers in a large duchenne muscular dystrophy cohort. Ann Neurol. 2016 Apr;79(4):535-47. doi: 10.1002/ana.24599. Epub 2016 Feb 19. PMID 26891991
- [Background] Forbes SC, Willcocks RJ, Triplett WT, Rooney WD, Lott DJ, Wang DJ, Pollaro J, Senesac CR, Daniels MJ, Finkel RS, Russman BS, Byrne BJ, Finanger EL, Tennekoon GI, Walter GA, Sweeney HL, Vandenborne K. Magnetic resonance imaging and spectroscopy assessment of lower extremity skeletal muscles in boys with Duchenne muscular dystrophy: a multicenter cross sectional study. PLoS One. 2014 Sep 9;9(9):e106435. doi: 10.1371/journal.pone.0106435. eCollection 2014. PMID 25203313
- [Background] Hurley DM, Williams ER, Cross JM, Riedinger BR, Meyer RA, Abela GS, Slade JM. Aerobic Exercise Improves Microvascular Function in Older Adults. Med Sci Sports Exerc. 2019 Apr;51(4):773-781. doi: 10.1249/MSS.0000000000001854. PMID 30489496
- [Background] Towse TF, Slade JM, Meyer RA. Effect of physical activity on MRI-measured blood oxygen level-dependent transients in skeletal muscle after brief contractions. J Appl Physiol (1985). 2005 Aug;99(2):715-22. doi: 10.1152/japplphysiol.00272.2005. Epub 2005 Mar 31. PMID 15802369
- [Background] Yoo JK, Pinto MM, Kim HK, Hwang CL, Lim J, Handberg EM, Christou DD. Sex impacts the flow-mediated dilation response to acute aerobic exercise in older adults. Exp Gerontol. 2017 May;91:57-63. doi: 10.1016/j.exger.2017.02.069. Epub 2017 Feb 16. PMID 28216412
- [Background] Kim SH, Choi YH, Cheon JE, Shin SM, Cho HH, Lee SM, You SK, Kim WS, Kim IO. Transient flow response after femoral artery catheterization for diagnostic neuroangiography in infants and children: Doppler US assessment of the ipsilateral femoral artery. Pediatr Radiol. 2015 Jan;45(1):86-93. doi: 10.1007/s00247-014-3071-4. Epub 2014 Jul 6. PMID 24997791
- [Background] Ely MR, Ratchford SM, La Salle DT, Trinity JD, Wray DW, Halliwill JR. Effect of histamine-receptor antagonism on leg blood flow during exercise. J Appl Physiol (1985). 2020 Jun 1;128(6):1626-1634. doi: 10.1152/japplphysiol.00689.2019. Epub 2020 May 14. PMID 32407239
- [Background] Porst H, Padma-Nathan H, Giuliano F, Anglin G, Varanese L, Rosen R. Efficacy of tadalafil for the treatment of erectile dysfunction at 24 and 36 hours after dosing: a randomized controlled trial. Urology. 2003 Jul;62(1):121-5; discussion 125-6. doi: 10.1016/s0090-4295(03)00359-5. PMID 12837435
- [Background] Taivassalo T, Jensen TD, Kennaway N, DiMauro S, Vissing J, Haller RG. The spectrum of exercise tolerance in mitochondrial myopathies: a study of 40 patients. Brain. 2003 Feb;126(Pt 2):413-23. doi: 10.1093/brain/awg028. PMID 12538407
- [Background] Miller NF, Alfano LN, Iammarino MA, Connolly AM, Moore-Clingenpeel M, Powers BR, Tsao CY, Waldrop MA, Flanigan KM, Mendell JR, Lowes LP. Natural History of Steroid-Treated Young Boys With Duchenne Muscular Dystrophy Using the NSAA, 100m, and Timed Functional Tests. Pediatr Neurol. 2020 Dec;113:15-20. doi: 10.1016/j.pediatrneurol.2020.08.013. Epub 2020 Aug 27. PMID 32979653
- [Background] Benitez-Porres J, Lopez-Fernandez I, Raya JF, Alvarez Carnero S, Alvero-Cruz JR, Alvarez Carnero E. Reliability and Validity of the PAQ-C Questionnaire to Assess Physical Activity in Children. J Sch Health. 2016 Sep;86(9):677-85. doi: 10.1111/josh.12418. PMID 27492937
- [Background] Gregor RJ, Broker JP, Ryan MM. The biomechanics of cycling. Exerc Sport Sci Rev. 1991;19:127-69. No abstract available. PMID 1936084
- [Background] Power LC, Gusso S, Hornung TS, Jefferies C, Derraik JGB, Hofman PL, O'Grady GL. Exercise Cardiac Magnetic Resonance Imaging in Boys With Duchenne Muscular Dystrophy Without Cardiac Disease. Pediatr Neurol. 2021 Apr;117:35-43. doi: 10.1016/j.pediatrneurol.2020.12.011. Epub 2020 Dec 30. PMID 33662889
- [Background] Laszlo G. Standardisation of lung function testing: helpful guidance from the ATS/ERS Task Force. Thorax. 2006 Sep;61(9):744-6. doi: 10.1136/thx.2006.061648. PMID 16936234
- [Background] McDonald CM, Widman L, Abresch RT, Walsh SA, Walsh DD. Utility of a step activity monitor for the measurement of daily ambulatory activity in children. Arch Phys Med Rehabil. 2005 Apr;86(4):793-801. doi: 10.1016/j.apmr.2004.10.011. PMID 15827934
- [Background] Washington SL 3rd, Shindel AW. A once-daily dose of tadalafil for erectile dysfunction: compliance and efficacy. Drug Des Devel Ther. 2010 Sep 7;4:159-71. doi: 10.2147/dddt.s9067. PMID 20856843
- [Background] Exercise Physiology In Special Populations. New York: Churchill Livingston Elsevier, 2008.
- [Background] Taivassalo T, Shoubridge EA, Chen J, Kennaway NG, DiMauro S, Arnold DL, Haller RG. Aerobic conditioning in patients with mitochondrial myopathies: physiological, biochemical, and genetic effects. Ann Neurol. 2001 Aug;50(2):133-41. doi: 10.1002/ana.1050. PMID 11506394
- [Background] Henrie AM, Nawarskas JJ, Anderson JR. Clinical utility of tadalafil in the treatment of pulmonary arterial hypertension: an evidence-based review. Core Evid. 2015 Nov 2;10:99-109. doi: 10.2147/CE.S58457. eCollection 2015. PMID 26587013
- [Background] Sabri MR, Beheshtian E. Comparison of the therapeutic and side effects of tadalafil and sildenafil in children and adolescents with pulmonary arterial hypertension. Pediatr Cardiol. 2014 Apr;35(4):699-704. doi: 10.1007/s00246-013-0840-z. Epub 2013 Nov 20. PMID 24253611
- [Background] Shiva A, Shiran M, Rafati M, Zamani H, Babazadeh K, Saeedi M, Ala S. Oral Tadalafil in Children with Pulmonary Arterial Hypertension. Drug Res (Stuttg). 2016 Jan;66(1):7-10. doi: 10.1055/s-0034-1395510. Epub 2015 Jan 22. PMID 25611962
- [Background] Takatsuki S, Calderbank M, Ivy DD. Initial experience with tadalafil in pediatric pulmonary arterial hypertension. Pediatr Cardiol. 2012 Jun;33(5):683-8. doi: 10.1007/s00246-012-0180-4. Epub 2012 Mar 9. PMID 22402804
- [Background] Yamazaki H, Kobayashi N, Taketsuna M, Tajima K, Suzuki N, Murakami M. Safety and effectiveness of tadalafil in pediatric patients with pulmonary arterial hypertension: a sub-group analysis based on Japan post-marketing surveillance. Curr Med Res Opin. 2017 Dec;33(12):2241-2249. doi: 10.1080/03007995.2017.1354832. Epub 2017 Jul 20. PMID 28699846
- [Background] Ferguson-Sells L, Velez de Mendizabal N, Li B, Small D. Population Pharmacokinetics of Tadalafil in Pediatric Patients with Pulmonary Arterial Hypertension: A Combined Adult/Pediatric Model. Clin Pharmacokinet. 2022 Feb;61(2):249-262. doi: 10.1007/s40262-021-01052-8. Epub 2021 Aug 11. PMID 34379314
- [Background] Martin EA, Barresi R, Byrne BJ, Tsimerinov EI, Scott BL, Walker AE, Gurudevan SV, Anene F, Elashoff RM, Thomas GD, Victor RG. Tadalafil alleviates muscle ischemia in patients with Becker muscular dystrophy. Sci Transl Med. 2012 Nov 28;4(162):162ra155. doi: 10.1126/scitranslmed.3004327. PMID 23197572